CLINICAL TRIAL: NCT01100710
Title: Relative Contribution of Age, Gender and Left Ventricular Mass as Quantified by Cardiac Magnetic Resonance Tomography to Detectable Levels of Cardiac Troponin T in a Healthy Reference Population Aged Below 70 Years
Brief Title: Age Gender Left Ventricular Mass and Cardiac Troponin T
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. med. E. Giannitsis, University Hospital Heidelberg
Other Study IDs: UHD
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2007-02

CONDITIONS: Heart Failure
Keywords: Age Gender left ventricular mass high sensitive Troponin T
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy volunteers

SUMMARY:
The purpose of this study is to determine the influence of functional or anatomic cardiac parameters, age and gender on high sensitivity cTnT (TnThs) levels in healthy individuals.

DETAILED DESCRIPTION:
We sought to investigate the relative contribution of functional or anatomic parameters as assessed by cardiac magnetic resonance tomography (cMRI, 1.5 Tesla), and clinical variables including increasing age and gender on high sensitivity cTnT (TnThs) levels in healthy individuals. Therefore we measured TnThs in serum samples of 120 healthy volunteers aged between 20 and 70 years. All individuals underwent cMRI including stress testing using dobutamine or adenosine.TnThs concentrations were related to cMRI and clinical findings. Partial correlation, as well as linear and hierarchical regression analyses were used to identify independent predictors and their relative contribution for prediction of TnThs values.

ELIGIBILITY:
Inclusion Criteria:

* agreement, age > 18 years, men and women

Exclusion Criteria:

* measurable heart disease, any chronic or acute disease, intake of meds, hypertension, Diabetes

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residents of Heidelberg and urban hinterland
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2007-03; Primary Completion 2007-03 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giannitsis, Prof., Principal Investigator
Locations (1):
- University Hospital of Heidelberg, Heidelberg, Baden-Würtemberg, Germany

REFERENCES:
- [Background] Apple FS, Smith SW, Pearce LA, Ler R, Murakami MM, Benoit MO, Levy C, Dumas C, Paul JL. Use of the bioMerieux VIDAS troponin I ultra assay for the diagnosis of myocardial infarction and detection of adverse events in patients presenting with symptoms suggestive of acute coronary syndrome. Clin Chim Acta. 2008 Apr;390(1-2):72-5. doi: 10.1016/j.cca.2007.12.016. Epub 2008 Jan 11. PMID 18230357